CLINICAL TRIAL: NCT01313910
Title: CCRC: A Pilot Project of the Treatment of HIV Enteropathy With ImmunoLin® Supplements
Brief Title: CCRC: A Project of the Treatment of HIV Enteropathy With ImmunoLin® Supplements
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Proliant Health & Biologicals (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 225193; 201118675 (Other: UC Davis)
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-05

CONDITIONS: HIV
Keywords: HIV; diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ImmunoLin® (Experimental): 8-week treatment course
  Interventions: Dietary Supplement: Immunolin®

INTERVENTIONS:
Dietary Supplement: Immunolin® — Immunolin® 500 mg capsules to be taken 5 capsules twice daily for eight weeks

SUMMARY:
The purpose of the study is to see if ImmunoLin® will reduce the frequency of bowel movements and gastrointestinal (GI) symptoms in HIV volunteers with persistent GI symptoms. The study will also examine the effect of ImmunoLin® on the bacteria in the gut and the immune system in gut tissue as well as in the blood.

ELIGIBILITY:
Inclusion Criteria:

* GI complaints consisting of at least 2 loose or watery stools per day or marked abdominal bloating that adversely effects activities of daily living (ADLs) or common social functioning for greater than 6 months, even though the symptomatology may wax and wane over that time period.
* Subjects should have had routine testing to exclude enteric pathogens.
* Subjects should have made an effort to identify food intolerance, especially lactose intolerance.
* Symptoms should be believed to be independent of ART or other medications known to have the potential to cause similar GI complaints; either because the symptoms predate initiation of the medications or shifts between different options for ART has had no appreciable effect on symptoms.
* Over the previous 6 months, alcohol use should be characterized as occasional with less than 1.5 ounces per day being the maximum estimated use (<2 beers or glasses of wine or 1 drink of hard liquor).
* Subjects will be greater than 18 years of age.
* Plasma HIV load should be suppressed to less than 400 cp/mL for at least four months, but there is no restriction on peripheral CD4+ T-cell count. Blips of <1000 cp/mL are allowed, provided that these are not associated with medication interruptions and that the pVL is undetectable before and after the observed blip.
* Subjects are willing to maintain a food and GI-symptom diary while receiving the ImmunoLin® supplement.
* Subjects should be willing to attempt to maintain a stable regimen of ART for the duration of the study unless indicated for patient safety.
* Subjects should be free of antibiotic use for at least 3-weeks prior to study entry except for chronic antibiotics used for prophylaxis according to SOC in HIV management. Usage of antibiotics during the course of the study will be assessed on a case by case basis by the study team.
* Subjects must be free of conditions which require chronic therapy that are known to alter the gut flora. Steroid use must be limited to intermittent topical preparations only which includes inhaled or dermatologic routes of application.

Exclusion Criteria:

* known unrelated causes for GI abnormalities.
* abnormal coagulation parameters (PT>1.2 ULN)
* thrombocytopenia (platelet count <50,000 within 6 weeks)
* contra-indications to upper endoscopy or conscious sedation
* anemia (> grade 1 [appendix D])
* aspirin, ibuprofen, warfarin or other agents that interfere with the coagulation cascade are prohibited within 1 week of endoscopy.
* positive pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M. Asmuth, MD, Principal Investigator — University of California, Davis Int Med: ID
Locations (1):
- UCD CTSC Clinical Research Center (CCRC), Mather, California, United States

REFERENCES:
- [Result] Asmuth DM, Ma ZM, Albanese A, Sandler NG, Devaraj S, Knight TH, Flynn NM, Yotter T, Garcia JC, Tsuchida E, Wu TT, Douek DC, Miller CJ. Oral serum-derived bovine immunoglobulin improves duodenal immune reconstitution and absorption function in patients with HIV enteropathy. AIDS. 2013 Sep 10;27(14):2207-17. doi: 10.1097/QAD.0b013e328362e54c. PMID 23660579

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with diagnosis of HIV enteropathy are eligible for enrollment.
Groups:
- ImmunoLin®: 2.5 grams twice daily for eight weeks
Period: Overall Study
Arm/Group | ImmunoLin®
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ImmunoLin®
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Bowel Movements Per Day
Description: self-reported bowel movement in diary
Time Frame: 8 weeks (56 days)
Measure: Median (Inter-Quartile Range); unit: bowel movements/day
Arm/Group | ImmunoLin®
Number analyzed (Participants) | 8
bowel movements/day
  baseline stool frequency | 5.8 [5 to 8.4]
  week-8 stool frequency | 2 [2 to 3.8]
Statistical Analysis 1: Comparison: ImmunoLin®; Wilcoxin-rank test used to determine decrease in bowel movements/day after 8 weeks of intervention; Test type: Superiority or Other; p = 0.008, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Frequency of Pro-inflammatory Bacterial Orders
Description: 16S rDNA sequencing for Bacteroidetes/Firmicutes ratio
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: ratio of Bacteroidetes/Firmicutes %
Arm/Group | ImmunoLin®
Number analyzed (Participants) | 8
ratio of Bacteroidetes/Firmicutes %
  baseline Bacteroidetes/Firmicutes ratio | 0.27 [0.20 to 0.54]
  week-8 Bacteroidetes/Firmicutes ratio | 0.55 [0.37 to 0.92]
Statistical Analysis 1: Comparison: ImmunoLin®; Test type: Superiority or Other; p = 0.11, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Measures of Gut Permeability
Description: five-hour disaccharide absorption test
Time Frame: 8 weeks
Measure: Mean (Inter-Quartile Range); unit: percentage absorption
Arm/Group | ImmunoLin®
Number analyzed (Participants) | 8
percentage absorption
  baseline permiability ratio | .024 [0 to .048]
  week-8 permeability ratio | 0.032 [0 to 0.047]
Statistical Analysis 1: Comparison: ImmunoLin®; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Systemic Immune Activation
Description: CD8+ T-cells with an activated phenotype (HLA-DR/CD38+ coexpression)
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: % CD8/HLA-DR/CD38+
Arm/Group | ImmunoLin®
Number analyzed (Participants) | 8
% CD8/HLA-DR/CD38+
  baseline CD8+ activation | 20.1 [17.8 to 27.9]
  week-8 CD8+ activation | 20.3 [17.8 to 29.2]

5. Secondary Outcome: Duodenal Immune Reconstitution
Description: changes in duodenal lamina propria CD3+/CD4+ density by immunohistochemistry
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: CD3+/CD4+ per mm^2 lamina propria
Arm/Group | ImmunoLin®
Number analyzed (Participants) | 8
CD3+/CD4+ per mm^2 lamina propria
  baseline duodenal CD3+/CD4+ cells | 213 [66 to 266]
  8 week duodenal CD3+/CD4+ cells | 322 [228 to 433]
Statistical Analysis 1: Comparison: ImmunoLin®; Test type: Superiority or Other; p = 0.016, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | ImmunoLin®
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
pilot open label study with eight subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No